CLINICAL TRIAL: NCT04547621
Title: The Combination of Hypofractionated Stereotactic Radiotherapy and Chemoradiotherapy Using Intensity-Modulated Radiotherapy for Newly Diagnosed Glioblastoma Multiforme: A Prospective, Single-Center, Single-Arm Phase II Clinical Trial
Brief Title: HSRT and IMRT Chemoradiotherapy for Newly Diagnosed GBM
Acronym: HSCK-010
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Enmin Wang, M.D., Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2020-791
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Glioma, Malignant
MeSH Terms: conditions — Glioma | interventions — Radiotherapy; Temozolomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- HSRT+IMRT+Temozolomide (Experimental): * Intensity-modulated radiotherapy 20Gy/10fx, 5 days a week for 2 weeks.
  * Hypofractionated stereotactic radiotherapy 30Gy/5fx, 5 days a week for 1 week.
  * Temozolomide once daily (75mg/m2/d) orally administered concurrently with radiotherapy.
  Interventions: Device: Radiation; Drug: Temozolomide

INTERVENTIONS:
Device: Radiation — Intensity-modulated radiotherapy 20Gy/10fx
Device: Radiation — Hypofractionated Stereotactic Radiotherapy 30Gy/5fx
Drug: Temozolomide — Temozolomide 75 mg/m2 concurrently administered with RT.

SUMMARY:
This study aims to evaluate the safety and effectiveness of the combination of 30Gy/5fx HSRT and 20Gy/10fx IMRT adjuvant therapy. The total biological effective dose (BED) of the PTV is 72 Gy in a ratio of alpha/beta ratio of 3, which equals to the conventional 60Gy/30fx treatment. This study can provide evidence for future non-inferiority phase III randomized controlled trials. The abbreviated course of radiotherapy can reduce the treatment time by half, benefit patients, and utilize the health resource.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years of age;
2. Karnofsky performance status (KPS) ≥ 60 within 14 days prior to registration;
3. Histopathologically proved diagnosis glioblastoma multiforme;
4. Underwent surgery, gross total resection or subtotal resection;
5. Estimated survival of at least 3 months;
6. Hgb > 90/gL; absolute neutrophil count (ANC) > 1.5×109/L, platelets > 80×109/L; Creatinine < 1.5 times the upper limit of laboratory normal value; Bilirubin < 2 times the upper limit of laboratory normal value; serum glutamate pyruvate transaminase (SGPT) or serum glutamate oxaloacetate transaminase (SGOT) < 3 times the upper limit of laboratory normal value;
7. Signed informed consent form;
8. Agreed to participate in the follow-up.

Exclusion Criteria:

1. Prior invasive malignancy unless disease free;
2. Received irradiation or other anti-tumor adjuvant therapies;
3. Brain stem disease or tumor greater than 6 cm in maximum diameter;
4. Prior therapy with an inhibitor of vascular endothelial growth factor (VEGF) or VEGFR;
5. Pregnancy or nursing mothers;
6. Participated in other trials after diagnosis;
7. Influence factors toward oral medications;
8. Patients with CTCAE5.0 grade 3+ bleeding within 4 weeks prior to registration;
9. Suffering from severe cardiovascular disease: myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmias (including men with QTc interval ≥ 450 ms, women ≥ 470 ms); according to NYHA criteria, grades III to IV Insufficient function, or cardiac color Doppler ultrasound examination indicates left ventricular ejection fraction (LVEF) <50%;
10. Long-term unhealed wounds or fractures;
11. History of organ transplantation;
12. Serious diseases that endanger patients' safety or affect patients' completion of research, according to the researchers' judgment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From the start of treatment to the date of death or the last follow-up, up to approximately 24 months
  Estimated using the Kaplan-Meier method

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From the start of treatment to the date of disease progression or death, up to approximately 24 months
  Estimated using the Kaplan-Meier method
Objective response rate (ORR) | Bimonthly up to intolerance the toxicity or progressive disease (PD), up to approximately 24 months
  ORR is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Assessment in Neuro-Oncology (RANO) prior to progression or any further therapy.
Quality of Life score (QoL) | Bimonthly up to intolerance the toxicity or PD, up to approximately 24 months
  European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) version 3.0
Cognitive function | Bimonthly up to intolerance the toxicity or PD, up to approximately 24 months
  Mini-Mental State Exam (MMSE, score range 0 to 30) to evaluate the cognitive function. Any score of 24 or more (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment.
Toxicity rate | Bimonthly up to intolerance the toxicity or PD, up to approximately 24 months
  Common Terminology Criteria for Adverse Events (CTCAE) 5.0 to assess the toxicity. Estimated using an exact binomial distribution together with 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Enmin Wang, MD, Principal Investigator — CyberKnife Center, Department of Neurosurgery, Huashan Hospital
Locations (1):
- CyberKnife Center, Department of Neurosurgery, Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Martinez-Carrillo M, Tovar-Martin I, Zurita-Herrera M, Del Moral-Avila R, Guerrero-Tejada R, Saura-Rojas E, Osorio-Ceballos JL, Arrebola-Moreno JP, Exposito-Hernandez J. Salvage radiosurgery for selected patients with recurrent malignant gliomas. Biomed Res Int. 2014;2014:657953. doi: 10.1155/2014/657953. Epub 2014 May 7. PMID 24895599
- [Background] Roa W, Kepka L, Kumar N, Sinaika V, Matiello J, Lomidze D, Hentati D, Guedes de Castro D, Dyttus-Cebulok K, Drodge S, Ghosh S, Jeremic B, Rosenblatt E, Fidarova E. International Atomic Energy Agency Randomized Phase III Study of Radiation Therapy in Elderly and/or Frail Patients With Newly Diagnosed Glioblastoma Multiforme. J Clin Oncol. 2015 Dec 10;33(35):4145-50. doi: 10.1200/JCO.2015.62.6606. Epub 2015 Sep 21. PMID 26392096
- [Derived] Guan Y, Pan M, Yang J, Lu Q, Han L, Liu Y, Li J, Zhu H, Gong X, Mei G, Liu X, Pan L, Dai J, Wang Y, Wang E, Wang X. A phase II open label, single arm study of hypofractionated stereotactic radiotherapy with chemoradiotherapy using intensity-modulated radiotherapy for newly diagnosed glioblastoma after surgery: the HSCK-010 trial protocol. BMC Cancer. 2022 Jul 29;22(1):827. doi: 10.1186/s12885-022-09914-5. PMID 35906549